CLINICAL TRIAL: NCT00622011
Title: Risperidone and Zotepine in the Treatment of Delirium
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: inadequate participant
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCH070906; CCH grant
Record Dates: First submitted 2008-01-31; First posted 2008-02-22 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Risperidone; zotepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): zotepine , start from 50mg/day then titrate according to individual case
  Interventions: Drug: Risperidone and Zotepine for delirium
- 2 (Active Comparator): Risperidone, start from 1mg/day
  Interventions: Drug: Risperidone and Zotepine for delirium

INTERVENTIONS:
Drug: Risperidone and Zotepine for delirium — try risperidone or zotepine in the treatment of delirium
  Other Names: risperidone( Risperdal), zotepine( Lodopine)

SUMMARY:
Delirium is an organic psychiatric syndrome characterized by fluctuating consciousness and impairment in perception, cognition and behavior. In hospitalized elderly, the prevalence of delirium ranges from 10% to 40%. If untreated, delirium is associated with significant morbidity and mortality. Treatment of delirium consists of identifying and managing underlying medical abnormalities and the associated psychiatric symptoms. Conventional antipsychotics have been the mainstay of treatment of agitation and psychosis associated with delirium; but their use is limited in terms of EPS side effects. Second-generation antipsychotic agents have been reported to have a lower incidence of extrapyramidal side effects and tardive dyskinesia which has resulted in their increased use in the treatment of delirious patients. However, there is still no consensus regarding standard pharmacologic treatment of this syndrome that takes use of second-generation antipsychotic agents into account.

Risperidone and zotepine have a lower incidence of EPS and are effective in treating disturbing psychotic behaviors. We hope to compare the efficacy and safety of risperidone and zotepine in the treatment of delirium and the correlation between the severity of delirium with autonomic dysfunction.

DETAILED DESCRIPTION:
Qualified inpatients will be enrolled and randomly given a flexible-dose regimen of Risperidone or Zotepine. Autonomic dysfunction is checked using analysis of heart rate variability before any active drug given. The initial starting dose of each drug is 1mg(risperidone) or 50 mg(zotepine) once a day. The dosage was increased depending on the status of delirium during the first 7 days and will be adjusted until patients are maximally stabilized or until intolerable adverse events necessitated cessation. Risperidone or zotepine will be tapered off in 10 days when patients are considered stable. No concomitant psychotropic medications will be used during the study except for lorazepam, which are given for severe agitation or insomnia . Patients are assessed by another rater blinded to active drug at the time of enrollment, the subsequent 12, 24,and then assessed daily until discharge. The study period is estimated to be around 12 months upon the designed number of subjects are reached.

ELIGIBILITY:
Inclusion Criteria:

* Patients may be included in the study if they meet all of the following criteria:DSM-IV-TR delirium (293.0 delirium due to general medical condition, 290.3 dementia with delirium 290.41, arteriosclerotic dementia with delirium 780.09delirium NOS. 292.8 substance-induced delirium( excluding alcohol and BZD)
* Age 18 to 85 year-old inpatients; either sex
* Patients are able to take Risperidone or Zotepine orally

Exclusion Criteria:

* Alcohol-induced delirium; delirium caused by seizures; Sedative, hypnotic or anxiolytic withdrawal delirium
* Patients with schizophrenia or bipolar disorder or being treated with antipsychotics
* Patients are mandatory to take parenteral treatments
* Patients are known to be allergic to Risperidone or Zotepine
* Women with pregnancy or during lactation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Delirium rating scale | 1/2 day, then every 24 hours

SECONDARY OUTCOMES:
MMSE, CGI, side effect profile, HRV | 12 hours, then every 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Chen Chang, M.D., Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan

REFERENCES:
- [Background] Boettger S, Breitbart W. Atypical antipsychotics in the management of delirium: a review of the empirical literature. Palliat Support Care. 2005 Sep;3(3):227-37. doi: 10.1017/s1478951505050352. PMID 16594462